CLINICAL TRIAL: NCT05709899
Title: Comparison of Ultrasound-guided Erector Spinae Plane Block and Transmuscular Quadratus Lumborum Block in Abdominal Cancer Surgeries.
Brief Title: Comparison of Ultrasound-guided Erector Spinae Plane Block and Transmuscular Quadratus Lumborum Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rana Ahmed Hamed Mohamed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: postoperative analgesia
Record Dates: First submitted 2022-10-27; First posted 2023-02-02 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Nerve Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I : Bilateral erector spinae plane block at L1 (Other): Ultrasound (US) will be used to identify the level of L1 after skin sterilization with the patient on the lateral position. A high frequency linear-array US transducer covered in a sterile sleeve will be placed in a longitudinal parasagittal orientation 3 cm lateral to the midline to identify the trapezius above, the rhomboid major in the middle, and the erector-spinae muscle on the bottom, and the transverse Processes with shimmering pleura in between. 2-3 ml of 2% lidocaine "depocaine HCL" will be infiltrated.16-G, 8-cm Tuohy needle will be then introduced medially in the plane of the US beam and directed towards the transverse process. Once the needle is underneath the anterior fascia of the erector spinae muscle. 20 ml of bupivacaine 0.25% "sunnypivacaine" will be injected in this potential space over five minutes. The injectate will be observed spreading underneath the ES muscle lifting the muscle of the transverse process. This will be repeated on the opposite side.
  Interventions: Other: nerve blocks
- Group II : Transmuscular quadratus lumborum block at L1 (Other): Patient will be positioned in left lateral to obtain appropriate view of QL. Aseptic precautions will be taken by wearing sterile gown and sterile drapes. By using Ultrasound MacroMaxx™ with linear probe (HFL38_10-5 MHz) covered with sterile plastic sheath SiteRite placed in the anterior axillary line to visualize the typical triple abdominal layers. Then, the probe will be placed in the midaxillary line and at this juncture the layers of abdominal layers will start to taper. When the probe will be placed in the posterior axillary line as per the posterior approach, sonoanatomy will show first the transversus abdominis disappearing then the internal oblique and external oblique forming aponeurosis and appearance of QL noticed. At the junction of the tapered ends of abdominal muscles and QL, a 21 g 100 mm SonoPlexStimu cannula needle will be inserted in plane. Under ultrasound guidance, in that space 20 mL of 0.25% bupivacaine "sunnypivacaine"will be injected separating the fascia.
  Interventions: Other: nerve blocks

INTERVENTIONS:
Other: nerve blocks — Comparison of ultrasound-guided erector spinae plane block and transmuscular quadratus lumborum block for postoperative analgesia in abdominal cancer surgeries.

SUMMARY:
The objective of this study is to compare the postoperative analgesic effect of bupivacaine injection via ultrasound-guided erector spinae block versus transmuscular quadratus lumborum block in patients undergoing abdominal cancer surgery

DETAILED DESCRIPTION:
Surgical trauma activates numerous receptors leading to severe postoperative pain. Therefore, effective pain management is a priority of care and a patient right .

Postoperative pain may cause tachycardia, hypertension, increased cardiac work, nausea, vomiting, ileus. Also if it is inadequately managed may lead to detrimental Cardiovascular effects, pulmonary dysfunction, immune system, neuro-endocrine and metabolic effects, gastrointestinal, urinary dysfunction, coagulation system , cognitive dysfunction and also have psychological, economic and social adverse effects Good postoperative analgesia can prevent morbidity associated with abdominal surgeries by allowing pain-free, early ambulation and decreasing the risks of long hospital stay, thromboembolism, and other poor outcomes.

Adequate pain treatment is an important component of modern perioperative care and essential for a fast recovery. Choosing the optimal analgesic modality remains a topic of debate especially in major abdominal surgeries.

Various techniques have been tried to replicate the analgesic efficacy of TEA. They include transversus abdominis plane analgesia (TAP), rectus sheath analgesia (RS), wound infusion analgesia (WI) and transmuscular quadratus lumborum (TQL) analgesia.

However each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for all open abdominal surgeries.

The ultrasound (US)-guided erector spinae plane block (ESPB) was initially described by Forero et al.It as a relatively new technique, originally described to manage thoracic pain when performed at the T5 vertebra level, but it has also been successfully used for abdominal analgesia when performed at T7 level.

ESPB gained wide attention as it is a faster procedure that carries a lower risk of hypotension, can be used in patients with coagulopathy, easy to perform, and requires less training.

ESPB provides extensive, potent unilateral analgesia, performed by local anesthetic injection in the plane between the erector spinae muscle and the TP. The local anesthetic diffuses into the paravertebral space through spaces between adjacent vertebrae and blocks both the dorsal and ventral rami of the thoracic spinal nerves.

Bilateral ESPB performed at low thoracic levels provides satisfactory analgesia for abdominal surgeries in case reports and series describing abdominal exploration, cesarean section, ventral hernia repair, and abdominoplasty.

As LA widely spreads cranially and caudally when ESPB is performed, we think that ESPB can effectively be used as an analgesic method for abdominal surgeries.

The ultrasound-guided (USG) quadratus lumborum block QLB was first described by Rafael Blanco in a presentation at ESRA 2007 at the XXVI Annual ESRA Congress in Valencia, Spain. Blanco described a potential space posterior to the abdominal wall muscles and lateral to the quadratus lumborum muscle (QL) where Local anesthetics (LA) can be injected. This technique provides analgesia after abdominal surgeries due to spread of LA from its lumbar deposition cranially into the thoracic paravertebral space (TPVS) where lateral and anterior cutaneous branches from Th7 to L1 nerves can be blocked. This was proved later by Carney et al. who found traces of contrast agent in the TPVS following the block.

Quadratus lumborum block (QLB) under ultrasound has been one of the interfascial plane blocks being popularized in regional anesthesia over the last few years given the vast number of indications in a variety of abdomino-pelvic surgeries in pediatrics and adults. In clinical studies, it also has been shown to have opioid sparing effects and prolonged post-operative analgesia than more conventional procedures like TAP blocks.

Several approaches have been described for QLB. Lateral QLB (or QLB-1) where local anesthetic is injected at the anterolateral border of the QL muscle. Posterior QLB (or QLB-2) where LA is injected at the junction of QL muscle with the transversalis fascia., Another novel approach is the transmuscular QLB (or QLB-3), where the needle is advanced through the QL muscle, penetrating the ventral proper fascia of the QL muscle and LA is finally injected between the QL muscle and Psoas Major (PM) muscle. It is thought that this approach (QLB-3) does not result in redundant antero-lateral spread of the LA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients subjected to abdominal cancer surgery.
2. The enrolled age will be from 18 years to 70 years.
3. ASA I-II and NYHA I-II.

Exclusion Criteria:

1. ASA physical status >II, and NYHA >II.
2. Patient refusal.
3. body mass index >40 kg/m2.
4. preoperative opioid consumption.
5. a local infection at the incision site.
6. a history of hematological disorders or coagulation abnormality.
7. previous abdominal surgeries, severe hepatic or renal impairment
8. Anomalies of vertebral column.
9. Pregnant women.
10. Hypersensitivity to any of used drugs.
11. chronic pain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia | First 48 hours after surgery.
  to assess pain intensity at rest and during pain-provoking movements (deep breathing, coughing, mobilization) measured by VAS pain score (a visual analog scale scored from 0 to 10 where 0 = no pain and 10 = the worst pain imaginable) during the first 48 hours postoperatively.

REFERENCES:
- [Background] Azari L, Santoso JT, Osborne SE. Optimal pain management in total abdominal hysterectomy. Obstet Gynecol Surv. 2013 Mar;68(3):215-27. doi: 10.1097/OGX.0b013e31827f5119. PMID 23945838
- [Background] Liu SS, Richman JM, Thirlby RC, Wu CL. Efficacy of continuous wound catheters delivering local anesthetic for postoperative analgesia: a quantitative and qualitative systematic review of randomized controlled trials. J Am Coll Surg. 2006 Dec;203(6):914-32. doi: 10.1016/j.jamcollsurg.2006.08.007. Epub 2006 Oct 25. No abstract available. PMID 17116561
- [Background] Restrepo-Garces CE, Chin KJ, Suarez P, Diaz A. Bilateral Continuous Erector Spinae Plane Block Contributes to Effective Postoperative Analgesia After Major Open Abdominal Surgery: A Case Report. A A Case Rep. 2017 Dec 1;9(11):319-321. doi: 10.1213/XAA.0000000000000605. PMID 28727597
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Ueshima H, Otake H. Similarities Between the Retrolaminar and Erector Spinae Plane Blocks. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):123-124. doi: 10.1097/AAP.0000000000000526. No abstract available. PMID 27997492
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Borglum J, Jensen K, Christensen AF, Hoegberg LC, Johansen SS, Lonnqvist PA, Jansen T. Distribution patterns, dermatomal anesthesia, and ropivacaine serum concentrations after bilateral dual transversus abdominis plane block. Reg Anesth Pain Med. 2012 May-Jun;37(3):294-301. doi: 10.1097/AAP.0b013e31824c20a9. PMID 22476239
- [Background] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Result] Yamak Altinpulluk E, Garcia Simon D, Fajardo-Perez M. Erector spinae plane block for analgesia after lower segment caesarean section: Case report. Rev Esp Anestesiol Reanim (Engl Ed). 2018 May;65(5):284-286. doi: 10.1016/j.redar.2017.11.006. Epub 2018 Jan 17. English, Spanish. PMID 29352577